CLINICAL TRIAL: NCT01943331
Title: Colonization and Infection in Critically Ill Patients: a Multicenter, Prospective, Observational Study in Intensive Care Units (ICUs) in China
Brief Title: Epidemiological Investigation of CRBSI, VAP, CAUTI in Chinese ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Department of critical care medicine, Zhongda Hospital, Southeast University, China
Other Study IDs: nosocomial infection in ICU
Record Dates: First submitted 2013-03-30; First posted 2013-09-16 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2013-04

CONDITIONS: Nosocomial Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients admitted to ICU

SUMMARY:
The current protocol desires to implement a large-multicenter observational study of hospital acquired infection in ICU in China. The study will generate data on generate data about the epidemiology current management of nosocomial infection.

DETAILED DESCRIPTION:
The objectives are as followings:

1. Obtain incidence of three major nosocomial infection in ICU, catheter related blood stream infection(CRBSI), catheter related urinary tract infection (CRUTI), and ventilator associated pneumonia (VAP).
2. Determine the epidemic of etiology and condition of management of three major nosocomial infection in ICU in China.

ELIGIBILITY:
Inclusion Criteria:all patients admitted into ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted into ICU are eligible for this study. All the infected patients were treated by the attending physician, and the choice and adjustment of antibiotic were in accordance with the recommendations of ATS guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
morbidity | one year
  the incidence rate of VAP, CRBSI,CAUTI of critical ill patients in Chinese ICU

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Xie, Principal Investigator — Department of Critical Care Medicine, Zhongda Hospital
Locations (1):
- Department of Critical Care , Zhong-da Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xie J, Yang Y, Huang Y, Kang Y, Xu Y, Ma X, Wang X, Liu J, Wu D, Tang Y, Qin B, Guan X, Li J, Yu K, Liu D, Yan J, Qiu H. The Current Epidemiological Landscape of Ventilator-associated Pneumonia in the Intensive Care Unit: A Multicenter Prospective Observational Study in China. Clin Infect Dis. 2018 Nov 13;67(suppl_2):S153-S161. doi: 10.1093/cid/ciy692. PMID 30423055